CLINICAL TRIAL: NCT06409390
Title: A Pilot Study of Sequential ("First Strike, Second Strike") Therapies, Modeled on Evolutionary Dynamics of Anthropocene Extinctions, for Hormone Positive Metastatic Breast Cancer
Brief Title: Sequential Therapies Modeled on Evolutionary Dynamics for Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22617
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; trastuzumab deruxtecan; sacituzumab govitecan; Capecitabine; Fulvestrant; ribociclib; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequential therapy (Experimental): In this study sequential therapies will be administered.
  Strike 1: Cytoxan/Taxotere/GM-CSF Strike 2: Sacituzumab govitecan or trastuzumab deruxtecan Strike 3: Capecitabine Strike 4: Fulvestrant + CDK 4/6 inhibitor (ribociclib or abemaciclib)
  Interventions: Drug: Taxotere; Drug: Cytoxan; Drug: Trastuzumab deruxtecan; Drug: Sacituzumab govitecan; Drug: Xeloda; Drug: Fulvestrant; Drug: Ribociclib; Drug: Abemaciclib

INTERVENTIONS:
Drug: Taxotere — 75 mg/m2 once every 21 days for 4 cycles
  Other Names: Docetaxel
Drug: Cytoxan — 600 mg/m2 once every 21 days for 4 cycles
  Other Names: Cyclophosphamide
Drug: Trastuzumab deruxtecan — 5.4 mg/kg once every 21 days for 5 cycles
  Other Names: Enhertu
Drug: Sacituzumab govitecan — 10 mg/kg on days 1 and 8 cycled every 21 days for 5 cycles
  Other Names: Trodelvy
Drug: Xeloda — 1000 mg/m2 orally twice daily for 14 days cycled every 21 days for 5 cycles
  Other Names: Capecitabine
Drug: Fulvestrant — 500 mg intramuscular (IM) on days 1, 15 and 28 of the first cycle followed by every 28 days for a total of 4 cycles
  Other Names: Faslodex
Drug: Ribociclib — 600 mg orally daily 21 days on, 7 days off
  Other Names: Kisqali
Drug: Abemaciclib — 150 mg by mouth twice daily
  Other Names: Verzenio

SUMMARY:
The purpose of the study is to test a treatment strategy with currently approved drugs to see if it is practical to administer the available drugs in a new way that researchers hope could be more effective in treating metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years or older
* Histologically or cytologically confirmed diagnosis of hormone positive HER2 negative metastatic breast cancer per ASCO/CAP criteria (Allison et al, 2020, Wolff et al, 2018), with diagnosis established through either a breast/axillary biopsy or biopsy of a metastatic lesion.
* Hormone positive MBC previously treated with endocrine therapy with either an aromatase inhibitor or Tamoxifen (alone or in combination with a CDK4/6 inhibitor).
* Elevated breast tumor markers which may include cancer antigen 15-3 (CA 15-3) levels above the institutional upper limit of normal (ULN) range of 0.0-31.0 U/mL, cancer antigen 27-29 (CA 27-29) (range <38 U/mL) and/or elevated Carcinoembryonic antigen (CEA) above institutional upper limit of normal (range 0.0 - 5.2 ng/mL).
* Presence of measurable disease on imaging via RECIST v1.1.
* ECOG performance status 0-1.
* Participants must have adequate organ and marrow function as defined in the protocol.
* A negative pregnancy test for pre-menopausal women of childbearing potential.
* Pre-menopausal women of childbearing potential who are sexually active with a male partner must agree to use adequate contraception prior to the study, for the duration of study participation.
* Inclusion of minorities: patients of all races and ethnic groups who meet the above inclusion and below exclusion criteria are eligible for this trial.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Ability to understand and the willingness to sign a written informed consent document or have a legally authorized representative sign on the participant's behalf.

Exclusion Criteria:

* Have previously received Fulvestrant for treatment of their breast cancer.
* History of allergic reactions attributed to the study drugs.
* Documented brain metastasis or active or newly diagnosed CNS metastases, including meningeal carcinomatosis, because systemic treatment would need to be paused for these patients.
* Treatment with any investigational compound within 30 days prior to the first dose of study drugs or during this study.
* Diagnosis or treatment for another systemic malignancy within 2 years before the first dose of study drugs, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Uncontrolled intercurrent illness including-but not limited to-ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with advanced, symptomatic visceral spread, that are at risk of life-threatening complications in the short term, including massive uncontrolled effusions (peritoneal, pleural, pericardial), pulmonary lymphangitis.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
* Active infection including tuberculosis, hepatitis B (known positive HBV surface antigen [HBsAg]), or hepatitis C (HCV). Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Participants with positive HCV antibody are eligible if polymerase chain reaction is negative for HCV RNA.
* Concurrent or prior use of immunosuppressive medication within 14 days before the first dose of study drugs, with the following exceptions: premedication with dexamethasone, intranasal, inhaled, topical or local steroid injections, systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or its equivalent; steroids as premedication for hypersensitivity reactions (e.g., premedication for iodinated contrast allergy before CT scan).
* Inability to comply with protocol requirements.
* Pregnant and/or breastfeeding women are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Sequential Therapy | Up to 18 months
  The proportion of patients able to complete the sequence of therapies by the conclusion of the trial.

SECONDARY OUTCOMES:
Safety and Tolerability | Up to 18 months
  The proportion of patients who experience adverse events or serious adverse events.
No Evidence of Disease (NED) | Up to 18 months
  The proportion of patients who are able to reach NED status by the conclusion of the trial will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Aixa Soyano, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States